CLINICAL TRIAL: NCT00887744
Title: A Multicenter, Post Marketing Clinical Follow-up Study to Evaluate the Safety and Effectiveness of the Minimally Invasive Device APERIUS® in Degenerative Lumbar Spinal Stenosis With Symptomatic Neurogenic Intermittent Claudication
Brief Title: Intermittent Neurogenic Claudication Treatment With APERIUS®
Acronym: INCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0001-AP
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Spinal Stenosis
Keywords: Degenerative Lumbar Spinal Stenosis; Neurogenic Intermittent Claudication; Interpinous Device; Percutaneous
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aperius Treatment Arm (Other): Single Arm
  Interventions: Device: Aperius® Percutaneous Interspinous Spacer

INTERVENTIONS:
Device: Aperius® Percutaneous Interspinous Spacer — Implantation of the Aperius® device
  Other Names: Aperius®

SUMMARY:
The primary purpose of the study is to measure the change in severity of symptoms and ability to function in every day activities in patients suffering from degenerative lumbar spinal stenosis after treatment with the Aperius® device.

DETAILED DESCRIPTION:
The Intermittent Neurogenic Claudication Treatment with Aperius® (INCA) trial was designed as a multicenter single arm post-marketing study to evaluate the safety and effectiveness of the Aperius® in patients with degenerative lumbar stenosis with symptomatic neurogenic intermittent claudication.

One hundred fifty six patients with a history of Degenerative lumbar spinal stenosis (Lumbar level L1 to L5) at one or maximum 2 levels with symptoms of neurogenic intermittent claudication with or without back pain were included. All patients were followed for 12 months with visits at 48 hours, 7 days, 6 weeks, 6 and 12 months.

Primary effectiveness endpoint was assessed as the mean percentage change from baseline in Zurich Claudication Questionnaire for Symptom Severity at 6 weeks. Other effectiveness outcomes were percentage change in Zurich Claudication Questionnaire scores (ZCQ), Quality of laife Questionnaire scores (called EuroQuol 5D or EQ-5D), Visual Analogue Scale (VAS) pain scores (back, leg and buttock groin pain), pain medication and changes in walking distance from baseline to follow-up. Procedure and device related Serious Adverse Events were assessed throughout the complete 12 month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* History of Degenerative Lumbar Spinal Stenosis (Lumbar spine level from L1 -L5), confirmed by Magnetic Resonance Imaging (MRI) at one or maximal two levels, with symptoms of intermittent neurogenic claudication.
* Leg / Buttock / Groin pain, with or without back pain, relieved by flexion. If back pain is also present, it must be partially relieved when flexed.
* Able to sit for 50 minutes without pain.
* Able to walk a distance of 20 meters without pain.
* Patient states availability for and willing to perform all follow -up examinations.
* Patient signed informed consent form.
* Adults (minimum 21 years of age).

Exclusion Criteria:

* Previous lumbar surgery.
* Unremitting pain (leg/buttock/groin/back) in any spinal position.
* Axial back pain without leg/buttock/groin pain.
* Significant lumbar instability at the affected level: spondylolisthesis greater than grade 1 on a scale from 1-4.
* Objective motor deficit.
* Significant peripheral neuropathy by nerve conduction velocity tests (peroneal and sural nerves) according to the investigator.
* Cauda equina syndrome, defined as neural compression causing neurogenic bowel (rectal incontinence) or bladder dysfunction (retention or incontinence).
* Spinal Stenosis with clinical symptoms at one or more levels outside the L1-L5 lumbar region.
* Severe symptomatic Spinal Stenosis requiring immediate surgical decompression,according to the investigator or lumbar spinal stenosis at more than 2 levels.
* Lumbar Spinal Stenosis, caused by tumors, metastasis or Paget's disease.
* Vascular claudication and severe peripheral vascular disease. (Diminished dorsalis pedis or tibial pulses) that limits walking.
* History of primary or secondary osteoporosis defined as a DXA scan (=dual energy x-ray absorptiometry) of the hip showing T-score (=the number of standard deviations above or below the mean for the patient's age, sex and ethnicity) of more than 2.5 standard deviation below the mean in the presence of one or more fragility fractures.
* Active systemic infection or local infection at the level to treat.
* Major Depression according to Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria.
* Dementia and/or inability to give informed consent.
* Unable to complete the study.
* Pregnancy and breastfeeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2006-11; Primary Completion 2009-05 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Wuelfert, Pharm., Study Director — Medtronic Spinal & Biologics
Locations (12):
- Belgium (6):
  - Hospital Campus Middelheim, Antwerp
  - Academic Hospital Sint-Jan Brugge-Oostende AV, Bruges
  - Park Léopold Hospital, Brussels
  - Notre Dame de Grace Hospital, Gosselies
  - University Hospital Tivoli, La Louvière
  - Hospital du Grand Hornu, Mons
- Germany (5):
  - Klinik und Poliklinik für Orthopädie (Hospital), Cologne
  - Gemeinschaftspraxis Königsallee (Privat Clinic), Düsseldorf
  - University Hospital Erlangen, Erlangen
  - Asklepios Hospital Lindenlohe, Schwandorf in Bayern
  - Orthopädische Fachklinik Schwarzach (Hospital), Schwarzach
- Woodend Hospital, Aberdeen, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient entered the study on November 20, 2006 and the last patient's last visit was on May 21, 2009 with a total study duration of 30 months.
Pre-assignment Details: Not applicable. Single arm study
Groups:
- Aperius® Treatment Arm: The targetted patient population -intended to be treated with the Aperius® Percutaneous Interspinous Spacer- is subjects with degenerative lumbar spinal stenosis with symptomatic neurogenic intermittent claudication.
Period: Overall Study
Arm/Group | Aperius® Treatment Arm
Started | 162 (162 patients signed an informed consent but only 157 patients were treated with the Aperius.)
Completed | 128
Not Completed | 34
Not completed — Adverse Event | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 18
Not completed — Various reasons | 9

BASELINE CHARACTERISTICS:
Groups:
- Aperius® Treatment Arm: The targetted patient population -intended to be treated with the Aperius® Percutaneous Interspinous Spacer- is subjects with degenerative lumbar spinal stenosis with symptomatic neurogenic intermittent claudication. The Aperius is a device will be inserted at day 0 (surgery date). Normally no additional manipulations are needed once the device(s) are inserted into the body.
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change in Symptom Severity at 6 Weeks Compared to Baseline, Using the Patient Completed Zurich Claudication Questionnaire for Symptom Severity
Description: This score is based on seven questions (overall pain,pain frequency,pain in the back,pain in the leg,numbness,weakness,and balanced disturbance.The first 6 categories are scored 1 to 5 (none,mild,moderate, severe,very severe). Balance disturbance is scored in a 1-3-5 scale (None,sometimes,often).The symptom severity scale score is the unweighted mean of all answered items (missing scores are discarded) in the questionnaire. Scoring range= 1-5.The change is calculated as the scores at the later timepoint minus the earlier timepoint expressed in terms of percentage.
Time Frame: From baseline up to 6 weeks follow-up
Population: Intention-To-Treat: the population of patients who underwent the minimally invasive procedure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Percent change | -29.7 (23.4)

2. Primary Outcome: The Proportion of Patients Experiencing a Procedure or Device Related Serious Adverse Events During the First 7 Days Starting at the Surgical Procedure
Description: Adverse events were to be summarized by proportion. All Adverse events occurring within the first 7 days after the surgical procedure were to be analyzed:
  * Day of the procedure until P+1 (where P refers to the day of the surgical procedure)
  * P+2 until P+7
Time Frame: Starting at the surgical procedure till 7 days post-operatively
Measure: Number; unit: Proportion of patients (%)
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Proportion of patients (%) | 3.8

3. Secondary Outcome: Mean Percentage Change in Symptom Severity at 12 Months Compared to Baseline, Using the Patient Completed Zurich Claudication Questionnaire for Symptom Severity
Description: The Zurich Claudication questionnaire - Symptom Severity score is based on seven questions (overall pain,pain frequency,pain in the back,pain in the leg,numbness,weakness,and balanced disturbance.The first 6 categories are scored 1 to 5 (none,mild,moderate, severe,very severe). Balance disturbance is scored in a 1-3-5 scale (None,sometimes,often).This score is the unweighted mean of all answered items (missing scores are discarded). Scoring range= 1-5.
  The change is calculated as the scores at the later timepoint minus the earlier timepoint expressed in terms of percentage.
Time Frame: From baseline up to 12 months follow up
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Percent Change | 26.7 (25.8)

4. Secondary Outcome: Mean Percentage Change in Physical Function at 12 Months Compared to Baseline, Using the Zurich Claudication Questionnaire
Description: The Zurich Claudication Questionnaire - Physical Function score is the unweighted mean of six physical function questions ranging from 1 to 4. The six Physical Function questions ask about walking distance and ability to walk for pleasure, for shopping, and for getting around the house or apartment and from bathroom to bedroom. If more than one item was missing, the scale score was also to be considered as missing. The possible range of this score is 1.0 to 4.0.
  The change is calculated as the scores at the later timepoint minus the earlier timepoint expressed in terms of percentage.
Time Frame: From baseline up to 12 months
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Percent Change | 25.3 (27.7)

5. Secondary Outcome: Mean Change in Quality of Life Score at 12 Months Compared to Baseline
Description: The quality of life scale covers five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels (no health problems,moderate health problems,extreme health problems). The distribution of the response of the patients in these five dimensions was to be studied.This descriptive system was converted into a weighted health state index with Min-max score = 0-100 and 100 as most optimal score. If one or more questions are left unanswered, the questionnaire is not scored.
Time Frame: From baseline up to 12 months follow up
Measure: Mean (Standard Deviation); unit: Scores on a scale (1-100)
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Scores on a scale (1-100) | 30 (31)

6. Secondary Outcome: Proportion of Patients Having Procedure and/or Device Related Events During the Complete 12 Month Follow-up Period.
Time Frame: From baseline up to 12 months follow up
Measure: Number; unit: Proportion of patients (%)
Arm/Group | Aperius® Treatment Arm
Number analyzed (Participants) | 157
Proportion of patients (%) | 7.6

ADVERSE EVENTS:
Time Frame: All Adverse events were gathered as from the moment the first patient entered the study on November 20, 2006 until the last patient's completed the last visit on May 21, 2009 with a total study duration of 30 months.
Description: All serious adverse device effects are listed below
Groups:
- ITT Analysis: Single group - Aperius
Arm/Group | ITT Analysis
Serious Adverse Events (participants affected / at risk) | 39/157
Other Adverse Events (participants affected / at risk) | 95/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Analysis (N=157)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 2 (2)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cholecystocholangitis (Hepatobiliary disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1) — Administrative site conditions
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2)
Muskuloskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal aneurysm (Renal and urinary disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Social stay hospitalization (Social circumstances) | 3 (3)
Spinal claudication (Nervous system disorders) | 6 (6)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Analysis (N=157)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (14)
Ataxia (Nervous system disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 40 (47)
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cystisis (Infections and infestations) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eye inflammation (Eye disorders) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Haematoma (Vascular disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Herpes Zoster (Infections and infestations) | 1 (1)
Hypoesthesia (Nervous system disorders) | 1 (1)
Hypogonadism (Endocrine disorders) | 1 (1)
Implant site swelling (General disorders) | 1 (1) — Administration site conditions
Incision site complication (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 2 (2)
Inflammation (General disorders) | 1 (1) — Administrative site conditions
Influenza (Infections and infestations) | 4 (4)
Influenza like illness (General disorders) | 2 (2) — Administration site conditions
Intervertbral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Lymphoedema (Vascular disorders) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 (32)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myocardial Ischaemia (Cardiac disorders) | 1 (1)
Nausea (Hepatobiliary disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nerve root lesion (Psychiatric disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2)
Oedema peripheral (Hepatobiliary disorders) | 1 (1) — and administration site conditions
Oral herpes (Infections and infestations) | 2 (2)
Osteitis (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (10)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1) — administration site conditions
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (31)
Paraesthesia (Nervous system disorders) | 6 (6)
Peripheral nerve lesion (Nervous system disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 4 (4)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Pyrexia (General disorders) | 3 (3) — administration site conditions
Radiation exposure (Injury, poisoning and procedural complications) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Sciatica (Nervous system disorders) | 5 (6)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensorimotor disorder (Nervous system disorders) | 1 (2)
Sensory disturbance (Nervous system disorders) | 3 (3)
Skeletal injury (Injury, poisoning and procedural complications) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Spinal claudication (Nervous system disorders) | 25 (26)
Spinal fracture (Injury, poisoning and procedural complications) | 3 (4)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator acknowledge that all information affecting or relating to Sponsor's products that is developed, discovered, or transmitted in connection with the study, including the multi-center data resulting from the study and any inventions or moral rights, shall belong to Sponsor, and nothing shall be construed to confer upon or grant to Institution or Investigator any right, title, or interest therein.